CLINICAL TRIAL: NCT02507362
Title: Adapted Fluence Settings for Corneal Collagen Cross-linking in Progressive Mild to Moderate Keratoconus Aged 18 to 30
Brief Title: Adapted Fluence Settings for Corneal Collagen Cross-linking in Mild to Moderate Progressive Keratoconus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ERC/S/9341
Record Dates: First submitted 2014-08-06; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Keratoconus
Keywords: keratoconus , corneal collagen cross-linking
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin; Subgingival Curettage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental (Experimental): Radiation: adjusted corneal collagen cross-linking (9mW/cm2 UV-A irradiation for 7 minutes after 30 mitunes of riboflavin instillation) riboflavin 0.1%: after mechanical epithelial removal riboflavin drop will be instilled every 5 minutes for 30 minutes and then instillation will be continued during irradiation epithelial debridement: corneal epithelium will be removed by a cottons swab
  Interventions: Radiation: adjusted corneal collagen cross-linking; Drug: riboflavin 0.1% combined with dextran 20 %; Procedure: epithelial debridement
- control (Active Comparator): radiation: accelerated corneal collagen cross-linking (9mW/cm2 UV-A irradiation for 10 minutes after 30 minutes of riboflavin instillation) riboflavin 0.1%: after mechanical epithelial removal riboflavin drop will be instilled every 5 minutes for 30 minutes and then instillation will be continued during irradiation epithelial debridement: corneal epithelium will be removed by a cottons swab
  Interventions: Radiation: accelerated corneal collagen cross-linking; Drug: riboflavin 0.1% combined with dextran 20 %; Procedure: epithelial debridement

INTERVENTIONS:
Radiation: adjusted corneal collagen cross-linking — UV-A irradiation for 7 minutes
  Arms: experimental
Radiation: accelerated corneal collagen cross-linking — UV-A irradiation for 10 minutes
  Arms: control
Drug: riboflavin 0.1% combined with dextran 20 % — after mechanical epithelial removal riboflavin drop will be instilled every 5 minutes for 30 minutes and then instillation will be continued during irradiation
Procedure: epithelial debridement — corneal epithelium will be removed by a cottons swab
  Other Names: epithelium removal

SUMMARY:
the purpose of this study is to compare the efficacy and safety of a new method of corneal cross-linking that uses UV-A irradiation intensity of 9mW/cm2 for 7 minutes to well-known Accelerated corneal cross-linking (9 mW/cm2 UV-A irradiation for 10 minutes)

DETAILED DESCRIPTION:
This study is a Prospective interventional clinical trial comparing two groups of mild to moderate progressive keratoconic patients; Control group will be treated with routine accelerated protocol of corneal cross-linking, while exposure time will be decreased in the experimental group.

we considered two groups of patients in our study:

* Group 1 (experimental): Exposure to 7 minutes at 9 mW/cm2 = 3.78 J/cm2
* Group 2 (controls): Exposure to 10 minutes at 9 mW/cm2 = 5.4 J/cm2

All demographic data of patients, their uncorrected distance visual acuity (UCDVA), corrected distance visual acuity (BCDVA), sphere and cylinder refraction, keratometry readings (k1 and k2) and other topographic parameters of the patients before the procedure and at every follow up visit will be recorded.

Corneal hysteresis and resistance factor will be checked by Ocular response analyzer before surgery and will be rechecked at 6 month follow up.

Intraoperative pain will also be recorded based on the visual analog scale (VAS + FACES pain scale) immediately after the completion of surgery.

Confocal microscopy will be used to evaluate changes in corneal stromal collagen fibers and keratocytes following cross-linking at 3 and 6 and 12 month post op period.

All procedures will be done by a single surgeon. We will use topical anesthesia by tetracaine followed by mechanical epithelial debridement at a radius of 9 millimeters. Then riboflavin 0.1% combined with dextran 20 % will be instilled every 3 minutes for 25 minutes. A short irrigation of the surface with BSS (to avoid a layer of riboflavin on the cornea during irradiation) will be performed. Corneal thickness will be determined by ultrasound pachymetry. If needed, hypoosmolar solution will be used to swell the cornea over 400 µm. If 400 µm cannot be reached, then irradiation will not be performed. Then we will irradiate the eye by the UV A light source 5cm away from the eye with a light intensity of 9 mW/cm2 for 10 minutes in control group and 7 minutes in experimental group and riboflavin will be instilled after 5 minutes for further in both groups, followed by a short irrigation of the surface with BSS (to avoid a layer of riboflavin on the cornea during irradiation).

After the procedure we will apply a bandage contact lens for 5- 7 days and will prescribe topical betamethasone every 6 hours for 2 weeks, tapered to TDS, BID and HS weekly for a total duration 5 weeks. A topical antibiotic drop (Oftaquix every 6 hours) will be used for the first week.

Patients will be followed up at day 1, day 6, 1 month, 3 months and 6 months and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate progressive KCN (Grade I and II) based on Amsler-krumeich classification; progression is defined as the old fashioned way in the lack of a consensus for more modern methods that is increase of > 1D of Kmax readings within 12 months
* Age> 18 y, and <35 years
* Kmax lower than 58 D
* Signing informed consent form

Exclusion Criteria:

* Any other ocular disease
* Corneal scar
* History of hydrops
* Any other ocular surgery including previous CCL, corneal inlay or keratorefractive surgery
* Inability to complete follow up schedule

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
keratometric values on pentacam measured by Javal keratometer | one year
best corrected visual acuity | one year
uncorrected distant visual acuity | one year

SECONDARY OUTCOMES:
clinical refraction | one year
endothelial cell count | one year

OTHER OUTCOMES:
corneal thickness | one year
corneal hysteresis | one year
corneal resistance factor | one year
intraoperative discomfort and pain | up to 1 hour
  Visual Analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Fateme Alipour, MD, Principal Investigator — Eye research center, Farabi eye hospital, Tehran university of medical science
Locations (1):
- Farabi eye hospital, Tehran, Tehran Province, Iran